CLINICAL TRIAL: NCT05606458
Title: The Effect of Multisensory Stimulation Applied by the Mother to Her Infant During the Heel Blood Collection Procedure on the Infant's Pain and Mother's State Anxiety: A Randomized Controlled Trial
Brief Title: The Effect of Multisensory Stimulation on Baby's Pain and Mother's Anxiety During Heel Blood Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Aysenur Akkaya Gul, Lecturer, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UludagUniversity/AKKAYAGUL
Record Dates: First submitted 2022-10-25; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Pain
Keywords: Neonatal; Heel Lance; Multisensory stimulation; Family Centered Care; NIPS; Sensorial Saturation(SS)
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The baby who met the inclusion and exclusion criteria underwent routine heel blood sampling at the hospital. First of all, the foot of the baby, who was taken to an open bed under a radiant heater, was warmed in the nurse's hand for one minute, the area where the baby's heel blood would be taken was determined, the baby's heel was wiped with 70% alcohol with the help of a sponge and waited for it to dry, then heel lance was performed. The procedure was completed after the relevant sections on the pre-prepared heel blood sheet were filled with blood. A light touch was provided if necessary for routine comfort of the infant for ethical reasons.
- İntervention Group (Experimental): Their mothers gave a multisensory stimulus to the newborns in the mother's room.
  1. Stimulus: Breast milk, breastfeeding (sense of taste)
  2. Stimulus : Maternal touch (sense of touch)
  3. Stimulus: Mother's voice (hearing sense)
  4. Stimulus: Maternal eye contact (sense of sight)
  5. Stimulus: Mother skin smell (sense of smell)
  Interventions: Behavioral: İntervention Group

INTERVENTIONS:
Behavioral: İntervention Group — Before the procedure, the baby was started to be breastfed (1st stimulus). The mother supported her baby's back and bottom with one hand. He started to touch by positioning the thumb of the other hand to prevent the baby's nose from being blocked, and the other fingers of the same hand to touch the baby's face (2nd stimulus). The mother started to talk to her baby with a gentle tone of voice, sometimes using sentences (lullaby, song, etc.) that she wanted to increase the volume of her voice (3rd stimulus). The mother was in the baby's sight (4th stimulus). Clothes were removed as much as possible for the smell of the mother's skin (5th stimulus). The baby's foot in the mother's arms was warmed in the nurse's hand for a minute. The area was determined, and the baby's heel was wiped with 70% alcohol. It was expected to dry. Heel piercing was performed while the stimuli continued. Heel blood was taken. When the evaluation period is complete, the process is over.
  Arms: İntervention Group

SUMMARY:
Newborn screening programs are preventive health services that have a significant place in public health programs in developed and developing countries worldwide. For these scans, heel blood is taken from the newborn, and the heel blood collection procedure applied for diagnostic purposes is one of the most common painful procedures applied to the newborn. Pharmacological and non-pharmacological pain management may be necessary to reduce and minimize pain during painful procedures in the neonatal intensive care unit. One of the non-pharmacological applications applied during acute procedural pain in the newborn is sensorial saturation, which consists of multisensory stimulation (sensitive touch, massage, auditory, visual, sense of taste, and smell). This study aimed to examine the effect of multisensory stimulation applied by the mother during the heel blood collection procedure in newborns on reducing pain and to evaluate the effects of family-centered practice on the state anxiety of mothers. This study was carried out as a randomized controlled, experimental study. Ethical approval was obtained before starting the study. In addition, written informed consent was obtained from the families of the newborns in the control and intervention groups. The study population consisted of newborns born in a hospital in Turkey between July 2019 and January 2020, and whose heel blood was taken for routine metabolic screening by the Ministry of Health. The sample group consisted of 80 randomly assigned newborns, 40 in the intervention group and 40 in the control group. Newborn mothers in the intervention group gave their babies multisensory stimulation(speech, touch, breastfeeding, eye contact, maternal skin odor) before, during, and after the procedure. The newborns in the control group underwent routine heel blood sampling in the baby room under a radiant heater. The Neonatal Infant Pain Scale (NIPS) was used for pain assessment. The NIPS score was evaluated by the researcher before the procedure, during the procedure, and 1 minute after the procedure. The State Anxiety Inventory was used to measure the mother's anxiety. The state of anxiety of the mothers in each group was evaluated before and after the procedure.

DETAILED DESCRIPTION:
Sensory stimuli can be easily realized with the active cooperation of the mother and, based on family-centered care, can help parents feel that they are playing an active role in their baby's care by being involved in their baby's care and can have positive effects on reducing the pain and stress of the baby during the heel blood collection process.As far as we know, there is no study in the literature investigating the effectiveness of multisensory stimulation applied by the mother during the heel blood collection procedure in reducing both the baby's pain and the mother's anxiety. It is thought that our study will provide new evidence to nursing care, that more than one sensory stimulus will be provided by the mother, will increase the baby's sense of confidence and reduce pain, contribute to the importance of family-centered care, and will be useful to support the results of the current study. This study aimed to examine the effect of multisensory stimulation applied by the mother during the heel blood collection procedure in newborns on reducing pain and to evaluate the effects of family-centered practice on the state anxiety of mothers.Before starting work, S.B.U. Ethical approval was obtained from the Süreyyapaşa Chest Diseases and Thoracic Surgery Clinical Research Ethics Committee. To start the research after the ethics committee's approval, T.C. Permissions were obtained from the Istanbul Provincial Health Directorate and the Istanbul Tuzla State Hospital management. In addition, written informed consent was obtained from the families of the newborns in the control and intervention groups. The research population consisted of all newborns born in Tuzla State Hospital in Turkey/Istanbul between July 2019 and January 2020 and whose infants were taken for routine metabolic screening by the Ministry of Health. The sample group consisted of 80 randomly assigned newborns, 40 in the intervention group and 40 in the control group. Randomization was provided according to the order of the procedure. The first newborn control group and the second newborn intervention group were formed. The newborns whose heel blood will be taken every day of the week during working hours continued from where they left off according to the order of the procedure. Before the procedure, the necessary materials were prepared, and the heel blood sheet information was filled in. The mothers of the babies whose heel blood was taken were informed about the heel blood screening and the research. The form containing the identification information of the baby and the mother was filled out. Before the procedure, the mother was asked to fill out the State Anxiety Scale (in both groups, the baby was with the mother). The newborns in the control group were taken to an open bed under a radiant heater, leaving the mother's side for routine heel blood collection applied in the hospital. First of all, the foot of the baby, who was taken to an open bed under a radiant heater, was warmed in the hands of the nurse for one minute, the area where the baby's heel blood would be taken was determined, the baby's heel was wiped with 70% alcohol with the help of a sponge and waited for it to dry, then heel lance was performed. The procedure was completed after the relevant sections on the pre-prepared heel blood sheet were filled with blood. A light touch was provided if necessary for the routine comfort of the baby for ethical reasons. The mothers of the babies whose heel blood was taken in the intervention group were informed about the steps of the procedure and the multisensory stimulation they would give to their babies (mother's voice, touching, breastfeeding, eye contact, mother's skin smell). The baby was started to be breastfed before the procedure and continued until the end of the evaluation period (1st stimulus). The mother supported her baby's back and bottom with one hand. He started to touch by positioning the thumb of the other hand to prevent the baby's nose from being blocked and the other fingers of the same hand to touch the baby's face (2nd stimulus). The mother started to talk with her baby in a gentle but firm tone, sometimes using sentences (words, lullabies, songs, etc.) that she wanted to increase the volume of her baby (3rd stimulus). Talking was started before the procedure and continued until the end of the evaluation period. The mother was in the baby's sight (4th stimulus). Clothes were removed as much as possible for the smell of the mother's skin (5th stimulus). After the baby's foot in the mother's lap was warmed in the nurse's hand for one minute, the area where the baby's heel blood would be taken was determined. After the baby's heel was wiped with 70% alcohol and a sponge and waited for it to dry, heel lance was performed. The procedure was completed after the relevant sections on the pre-prepared heel blood sheet were filled with blood. If the baby stopped sucking at any time during the procedure, the baby was placed back on the breast and the procedure continued from where it had left off. In the study, the data of the baby and the mother was prepared by the researcher mother's age, mother's occupation, gestational week of the baby, birth weight, gender, mode of delivery, etc.), the "Neonatal Infant Pain Scale (NIPS)" scale, which will be used in the assessment of the baby's pain, and the questionnaire form of the State Anxiety Scale to measure the mother's anxiety was used. NIPS score was evaluated by the researcher before the procedure, during the procedure, and 1 minute after the procedure. The State Anxiety Scale was administered to the mother before and after the procedure. The researcher calculated state anxiety scale scores.

ELIGIBILITY:
Inclusion Criteria:

* Being a term baby with a gestational age of 38-42 GH
* The birth weight of 2500 g or more
* Having a baby for whom only heel blood sampling will be performed
* Babies with a 5th-minute Apgar score of 7 and above
* Having a baby who did not receive any painful stimuli until 30 minutes before the intervention
* The criteria for the parent's willingness to participate in the study are sought.

Exclusion Criteria:

* Babies receiving muscle relaxants, analgesics, and sedation will not be included in the study.
* Voluntary refusal of parents to take heel blood

Ages: 38 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS) | Pre-procedure.
  The Neonatal Infant Pain Scale (NIPS) was used for pain assessment. The primary outcome was the pain score assessed with the NIPS scale, a validated and widely used tool to measure procedural pain in infants. NIPS is a measurement tool that includes five behavioral groupings (facial expression, crying, movements of arms and legs, state of alertness) and one physiological parameter (respiration pattern). Of the indicators, only crying is scored between 0 and 2, while the other indicators are scored as 0 or 1. Evaluation results in a possible total score between 0 and 7. A high score indicates an increase in the severity of pain. NIPS was evaluated before the procedure, during the procedure, and at the 1st minute after the procedure.
Neonatal Infant Pain Scale (NIPS) | During the procedure
  The Neonatal Infant Pain Scale (NIPS) was used for pain assessment. The primary outcome was the pain score assessed with the NIPS scale, a validated and widely used tool to measure procedural pain in infants. NIPS is a measurement tool that includes five behavioral groupings (facial expression, crying, movements of arms and legs, state of alertness) and one physiological parameter (respiration pattern). Of the indicators, only crying is scored between 0 and 2, while the other indicators are scored as 0 or 1. Evaluation results in a possible total score between 0 and 7. A high score indicates an increase in the severity of pain. NIPS was evaluated before the procedure, during the procedure, and at the 1st minute after the procedure.
Neonatal Infant Pain Scale (NIPS) | 1st minute after the procedure.
  The Neonatal Infant Pain Scale (NIPS) was used for pain assessment. The primary outcome was the pain score assessed with the NIPS scale, a validated and widely used tool to measure procedural pain in infants. NIPS is a measurement tool that includes five behavioral groupings (facial expression, crying, movements of arms and legs, state of alertness) and one physiological parameter (respiration pattern). Of the indicators, only crying is scored between 0 and 2, while the other indicators are scored as 0 or 1. Evaluation results in a possible total score between 0 and 7. A high score indicates an increase in the severity of pain. NIPS was evaluated before the procedure, during the procedure, and at the 1st minute after the procedure.
State-Trait Anxiety Scale | Pre-procedure
  The State-Trait Anxiety Inventory consists of two separate forms containing a total of 40 items. The State Anxiety Scale consists of 20 questions. Scoring the State Anxiety Inventory; According to the severity of the emotions, they are answered as (1) none, (2) a little, (3) a lot, and (4) completely. There are direct (straight) and reversed statements in the scales. Direct statements are negative emotions. Inverted expressions are positive emotions. The State Anxiety Scale has ten reversed statements (items 1, 2, 5, 8, 10, 11, 15, 16, 19, and, 20). Total score; It is found by subtracting the total score of positive statements from the total score of negative statements and adding 50, which is the constant value for this scale. Total score: "0-19 points" are considered as no anxiety, "20-39 points" as mild anxiety, "40-59 points" as moderate anxiety, "60-79 points" as severe anxiety, and "80 and above" as panic.
State-Trait Anxiety Scale | İmmediately after the procedure
  The State-Trait Anxiety Inventory consists of two separate forms containing a total of 40 items. The State Anxiety Scale consists of 20 questions. Scoring the State Anxiety Inventory; According to the severity of the emotions, they are answered as (1) none, (2) a little, (3) a lot, and (4) completely. There are direct (straight) and reversed statements in the scales. Direct statements are negative emotions. Inverted expressions are positive emotions. The State Anxiety Scale has ten reversed statements (items 1, 2, 5, 8, 10, 11, 15, 16, 19, and, 20). Total score; It is found by subtracting the total score of positive statements from the total score of negative statements and adding 50, which is the constant value for this scale. Total score: "0-19 points" are considered as no anxiety, "20-39 points" as mild anxiety, "40-59 points" as moderate anxiety, "60-79 points" as severe anxiety, and "80 and above" as panic.

CONTACTS AND LOCATIONS:
Locations (1):
- Uludag University, Bursa, Nilufer, Turkey (Türkiye)

REFERENCES:
- [Derived] Akkaya-Gul A, Ozyazicioglu N, Celikboya-Kabadayi E. Multisensory stimulation by mothers: impact on neonatal pain and maternal anxiety during heel blood collection: a randomized controlled trial. J Perinatol. 2025 Oct 6. doi: 10.1038/s41372-025-02436-5. Online ahead of print. PMID 41053317